CLINICAL TRIAL: NCT04986163
Title: Randomized Controlled Trial for Intraoperative Nociception Monitoring with Medstorm, Medasense and Anspec-pro During Total Intravenous Anesthesia (TIVA) Using Propofol and Remifentanil
Brief Title: Intraoperative Nociception Monitoring with Medstorm, Medasense and Anspec-pro During Total Intravenous Anesthesia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical issues
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BC-08020
Record Dates: First submitted 2021-05-25; First posted 2021-08-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pain Measurement

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The results of the pain monitors are masked for the investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- non-invasive analgesia monitoring with ANSPEC-PRO monitor and MEDASENSE monitor (Active Comparator): non-invasive analgesia monitoring with ANSPEC-PRO monitor and MEDASENSE monitor: the monitoring will be done in different periods. In each period the two monitors will monitoring the pain in a serial way. Period 1: awake patient, Period 2: sedated patient with propofol, Period 3 : monitoring during standardized pain stimulus; Period 4: monitoring during surgery
  Interventions: Device: Non-invasive analgesia monitoring with ANSPEC-PRO monitor and MEDASENSE monitor
- non-invasive analgesia monitoring with ANSPEC-PRO monitor and MEDSTORM monitor (Active Comparator): non invasive analgesia monitoring with ANSPEC-PRO and MEDSTORM the monitoring will be done in different periods. In each period the two monitors will monitoring the pain in a serial way. Period 1: awake patient, Period 2: sedated patient with propofol, Period 3 : monitoring during standardized pain stimulus; Period 4: monitoring during surgery
  Interventions: Device: Non-invasive analgesia monitoring with ANSPEC-PRO monitor and MEDSTORM monitor
- non-invasive analgesia monitoring with MEDSTORM and MEDASENSE (Active Comparator): non-invasive analgesia monitoring with MEDSTORM and MEDASENSE the monitoring will be done in different periods. In each period the two monitors will monitoring the pain in a serial way. Period 1: awake patient, Period 2: sedated patient with propofol, Period 3 : monitoring during standardized pain stimulus; Period 4: monitoring during surgery
  Interventions: Device: Non-invasive analgesia monitoring with MEDSTORM monitor and MEDASENSE monitor

INTERVENTIONS:
Device: Non-invasive analgesia monitoring with ANSPEC-PRO monitor and MEDSTORM monitor — The patients are monitored with two monitors under anesthesia: one monitor attached to the left hand and one monitor to the right hand. When one monitor is connected to the patient, the other monitor will be disconnected. The first monitor is ANSPEC and the second monitor used is MEDSTORM.
  Arms: non-invasive analgesia monitoring with ANSPEC-PRO monitor and MEDSTORM monitor
Device: Non-invasive analgesia monitoring with ANSPEC-PRO monitor and MEDASENSE monitor — The patients are monitored with two monitors under anesthesia: one monitor attached to the left hand and one monitor to the right hand. When one monitor is connected to the patient, the other monitor will be disconnected. The first monitor is ANSPEC-PRO and the second monitor used is MEDASENSE.
  Arms: non-invasive analgesia monitoring with ANSPEC-PRO monitor and MEDASENSE monitor
Device: Non-invasive analgesia monitoring with MEDSTORM monitor and MEDASENSE monitor — The patients are monitored with two monitors under anesthesia: one monitor attached to the left hand and one monitor to the right hand. When one monitor is connected to the patient, the other monitor will be disconnected. The first monitor is MEDSTORM and the second monitor used is MEDASENSE.
  Arms: non-invasive analgesia monitoring with MEDSTORM and MEDASENSE

SUMMARY:
The randomized controlled trial study aims to validate a new pain monitor during general anesthesia by comparing the new ANSPEC-PRO monitor (non-CE marked) with already CE-marked pain monitors (Medstorm and Medasense). One hundred and eighty patients will be randomized into six groups, wherein each group has 30 patients. Patients preparing for a surgical operation under general anesthesia will be included to be monitored for pain during surgery procedure, while the standard monitoring, medication, and standard care will not be disturbed.

Pain monitoring is done with the ANSPEC-PRO, MEDASENSE, or MEDSTORM in the operation room, before and during general anesthesia: the pain monitor will record data continuously, while the following will be recorded in parallel: blood pressure, heart rate, saturation, CO2, O2 end-tidal concentrations, electromyogram, signal quality, the given amount of analgesics and hypnotics, and TOF (train-of-four).

DETAILED DESCRIPTION:
Primary Objective: Validation of ANSPEC-PRO as pain monitor during general anesthesia.

Secondary Objectives

* Evaluation of quality of monitoring ANSPEC-PRO compared with other pain monitors (Medasense and Medstorm);
* Evaluation of the correlation between measurements of pain monitors (ANSPEC-PRO, Medstorm and Medasense) and the level of analgesia represented as TCI infusion of Remifentanil;
* To determine the most suitable device for the development of a MIMO pharmacodynamic interaction model of Propofol and Remifentanil for use in closed- loop drug-delivery systems for anesthesia;
* Evaluation of the interaction between analgesics and hypnotics measured by ANSPEC-PRO and BIS/Neurowave.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years and younger than 80 years
2. Patients able to comprehend, sign, and date the written informed consent document to participate in the clinical trial.
3. ASA Class I, II, III classified by the anesthesiologist.
4. Patients planned for a surgical procedure under general anesthesia.

Exclusion Criteria:

1. Patients having epidural analgesia infused by a pain pump during the operation.
2. Patients with chronic pain or getting medication used for chronic pain, like anti-epileptics, antidepressants, opioids.
3. Pregnant women (asked at the patient before the operation)
4. Patients with electrically sensitive life support systems (e.g. implanted pacemaker, defibrillator)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Registration of pain monitor output during surgery under general anesthesia | during general anesthesia for surgery
  validation of the pain monitor during aensthesia

CONTACTS AND LOCATIONS:
Overall Officials: Martine Neckebreoek, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publications are to be shared with UGent, Research Group on Dynamical Systems and Control, represented by prof. dr. Clara Ionescu.
Supporting Information: Study Protocol, CSR
Time Frame: The data will become available from the beginning of the study.
Access Criteria: All information will be available at martine.neckebroek@ugent.be (principal investigator)